CLINICAL TRIAL: NCT03303495
Title: A Multinational, Randomized, Phase III Study of FOLFIRI With/Without Bevacizumab Versus Irinotecan With/Without Bevacizumab As Second-line Therapy in Patients With Metastatic Colorectal Cancer
Brief Title: A Study of 2nd-line FOLFIRI ± Bevacizumab vs. Irinotecan ± Bevacizumab in mCRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor and President, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHANGE
Record Dates: First submitted 2017-09-23; First posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms
Keywords: FOLFIRI; CPT-11; Bevacizumab; 2nd-line metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms | interventions — Bevacizumab; Irinotecan; Fluorouracil; Leucovorin

ARMS (2):
- FOLFIRI +/- Bevacizumab (Experimental): Bevacizumab 5 mg/kg IV 90-30 min Day 1; CPT-11 180 mg/m2 IV 90 min Day 1; l-LV (dl-LV) 200 mg/m2 (400 mg/m2) IV 120 min Day 1; 5-FU - bolus 400 mg/m2 IV bolus Day 1; 5-FU - infusional 2400 mg/m2 IV continuous (46 hours) Day 1 - 3
  Interventions: Biological: Bevacizumab; Drug: CPT-11; Drug: 5-FU Bolus; Drug: 5-FU Infusion; Drug: l-LV (dl-LV)
- CPT-11 +/- Bevacizumab (Experimental): Bevacizumab 5 mg/kg IV 90-30 min Day 1; CPT-11 180 mg/m2 IV 90 min Day 1
  Interventions: Biological: Bevacizumab; Drug: CPT-11

INTERVENTIONS:
Biological: Bevacizumab — 5 mg/kg intravenously administered over 90 minutes (can be reduced to 30 minutes at the minimum) on day 1 of a 2-week cycle.
  Other Names: Avastin
Drug: CPT-11 — 180 mg/m2 intravenously administered over 90 minutes on day 1 of a 2-week cycle
  Other Names: Irinotecan
Drug: 5-FU Bolus — 400 mg/m2 intravenous bolus on day 1 of a 2-week cycle.
  Other Names: fluorouracil
  Arms: FOLFIRI +/- Bevacizumab
Drug: 5-FU Infusion — 2400 mg/m2 continuous infusion over 46 hours on day 1 and 2 of a 2-week cycle.
  Other Names: fluorouracil
  Arms: FOLFIRI +/- Bevacizumab
Drug: l-LV (dl-LV) — 200 (dl-LV: 400) mg/m2 intravenously administered over 120 minutes on day 1 of a 2-week cycle.
  Other Names: Leucovorin
  Arms: FOLFIRI +/- Bevacizumab

SUMMARY:
The primary purpose of this study is to determine the non-inferiority of overall survival FOLFIRI with or without Bevacizumab compared with Irinotecan (CPT-11) with or without Bevacizumab as Second-line therapy in Patient with Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
Primary endpoint: Overall survival (OS), Secondary endpoints: Progression-free survival (PFS), Time to treatment failure (TTF), Overall response rate (ORR),Disease Control Rate (DCR), Safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed inoperable colorectal adenocarcinoma excluding vermiform appendix cancer and anal canal cancer.
2. Age ≥18 years at the time of informed consent
3. ECOG performance status (PS) of 0-2
4. Written informed consent prior to study-specific screening procedures
5. Life expectancy of at least 90 days
6. Withdrawal from first-line chemotherapy (regardless of containing molecular-targeted drugs) for metastatic colorectal cancer due to intolerable toxicity or progressive disease, or relapse within 180 days after the last dose of adjuvant chemotherapy.
7. Adequate organ function according to following laboratory values obtained within 14 days before enrolment (excluding patients who received blood transfusions or hematopoietic growth factors within 14 days before the laboratory test) Neutrophil count: ≥1500/mm3 Platelet count: ≥10.0 x 104/mm3 Hemoglobin: ≥9.0 g/dL Total bilirubin: ≤1.5 mg/dL AST, ALT: ≤100 IU/L (≤200 IU/I if liver metastases present) Serum creatinine: ≤1.5 mg/dL

Exclusion Criteria:

1. History of other malignancy with a disease-free interval <5 years (other than curatively treated cutaneous basal cell carcinoma, curatively treated carcinoma in situ of the cervix, and gastroenterological cancer confirmed to be cured by endoscopic mucosal resection)
2. With massive pleural effusion or ascites requiring intervention
3. Radiological evidence of brain tumor or brain metastases
4. Active infection including hepatitis
5. Any of the following complication:

   i) Gastrointestinal bleeding or gastrointestinal obstruction (including paralytic ileus) ii) Symptomatic heart disease (including unstable angina, myocardial infarction, and heart failure) iii) Interstitial pneumonia or pulmonary fibrosis iv) Uncontrolled diabetes mellitus v) Uncontrolled diarrhea (that interferes with daily activities despite adequate therapy)
6. Any of the following medical history:

   Myocardial infarction: History of one episode within one year before enrollment or two or more lifetime episodes i) Serious hypersensitivity to any of the study drugs ii) History of adverse reaction to fluoropyrimidines suggesting dihydropyrimidine dehydrogenase (DPD) deficiency
7. Previous treatment with irinotecan hydrochloride
8. Current treatment with atazanavir sulfate
9. Previous treatment with tegafur, gimeracil, and oteracil potassium within seven days before enrollment
10. Pregnant or lactating females, and males and females unwilling to use contraception
11. Requires continuous treatment with systemic steroids
12. Psychiatric disability that would preclude study compliance
13. Otherwise determined by the investigator to be unsuitable for participation in the study
14. Concurrent gastrointestinal perforation or history of gastrointestinal perforation with 1 year before enrollment
15. History of pulmonary hemorrhage/hemoptysis ≥ Grade 2 (defined as bright red blood of at least 2.5mL) within 1 month prior to enrollment.
16. History of laparotomy, thoracotomy, or intestinal resection within 28 days before enrollment
17. Unhealed wound (except suture wounds from implantation of a central venous port), gastrointestinal ulcer, or traumatic fracture
18. Current or recent (within 1 year) thromboembolism or cerebrovascular disease
19. Currently receiving or requires anticoagulation therapy (> 325 mg/day of aspirin)
20. Bleeding diathesis, coagulopathy, or coagulation factor abnormality (INR ≥1.5 within 14 days before enrollment)
21. Uncontrolled hypertension
22. Urine dipstick for proteinuria >+2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2011-11-14 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Assessed until 1.5 years after the last patient enrolment
  Time from the date of enrollment to death from any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Assessed until 1.5 years after the last patient enrolment
  Time from the date of enrollment to the earlier of the date of confirmed progression or death from any cause.
Time to treatment failure (TTF) | Assessed until 1.5 years after the last patient enrolment
  Time from the date of enrollment to the earlier of the date of confirmed progression, death from any cause, or discontinuation of protocol treatment.
Overall Response Rate (ORR) | Assessed at 6, 12 week and thereafter every 8 weeks, from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks
  Proportion of eligible patients with measurable lesions with a best overall response of CR or PR assessed by the attending physician.
Disease Control Rate (DCR) | Assessed at 6, 12 week and thereafter every 8 weeks, from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks
  Proportion of best overall response of CR, PR, or SD assessed by the attending physician.
Incidence of Adverse Events (Adverse Reactions) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks
  The incidence of worst-grade adverse events (toxicities) on study as graded by NCI-CTCAE v 4.0 will be determined by treatment arm in all treated patients for the following events.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol